CLINICAL TRIAL: NCT04112277
Title: Observational Prospective Study of Opiate-free Anesthesia for Anterior Total Hip Replacement
Acronym: ASOPHA
Status: Completed | Type: Observational
Sponsor: Hôpital Privé Sévigné (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-A03393-52
Record Dates: First submitted 2019-09-30; First posted 2019-10-02 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Rehabilitation; Analgesia; Anesthesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Cumulative morphine consumption — morphine equivalent [mg] 24 hours after the procedure

SUMMARY:
Opioid-free anesthesia (ATO) is a multimodal anaesthesia combining different analgesic and anesthetic modalities thus excluding opiates as an intraoperative. Recent studies have found a benefit from the ATO on postoperative rehabilitation and reduced length of hospitalization.

Periarticular infiltration with a local anesthetic is one of the measures proposed in OFA during the PTH.

PTH remains a painful procedure and the occurrence of morphinic-related side effects in sometimes elderly patients is often observed.

The main objective of this study is to assess the feasibility of ATO in anterior hip replacement under general anesthesia with the primary endpoint of morphine consumption measured 24 hours after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and 85
* ASA (American Society of Anesthesiology) I-III
* Total Hip Prosthesis programmed anteriorly
* Prior obtaining free and informed written consent .Affiliation or beneficiary of a social security scheme. Patients affiliated with or beneficiaries of a social security plan and not included in another trial.

Exclusion Criteria:

* Pregnant women or breastfeeding Spinal anesthesia Patient on long-term opiate Body Mass Index (BMI) - 20 or 45kg/m2 Incomprehension of the ENS scale Unaccompanied cardiac conduction disorder, Adam-Stokes syndrome Preoperative Spontaneous Cardiac Frequency - 40 beats/min Left ventricle ejection fraction - 40% Unpaired sleep apnea syndrome (OSA) Adult incompetent, adults under guardianship or curatorial or deprived of liberty Allergy to one of the protocol products or their excipients: levobupivacaine, paracetamol, pregabalin, ketoprofen, dexmedetomidine Paracetamol-specific contraindication: hepatocellular deficiency Ketoprofen-specific contraindications: creatinine clearance - 60ml/min, ATCD of perforated peptic ulcer, heart failure, progressive hemorrhage, asthma associated with ketoprofen use Contraindications to nefopam: symptomatic prostate disorders, angle-closing glaucoma, epilepsy Participation in another clinical study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with ASA (American Society of Anesthesiology) I-III for whom a total Hip Prosthesis is programmed anteriorly (Hueler Method).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-02-25 (Actual); Study Completion 2020-02-25 (Actual)

PRIMARY OUTCOMES:
Cumulative morphine consumption | 24 hours after the procedure
  morphine equivalent [mg]

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Privé Sévigné, Cesson-Sévigné, France